CLINICAL TRIAL: NCT01358435
Title: Randomized,Single Center,Double Blind,Two-period,Crossover Glucose Clamp Trial Study to Test Bioequivalence Between Two Recombinant Human Mixed Insulins-Wockhardt's Human/Isophane Susp 30IU/ml/70IU/ml With Novolin70/30, in Healthy Subjects
Brief Title: Comparative Wockhardt's Glucose Clamp Study-Human Isophane Susp 30IU/ml/70IU/ml With Novolin70/30, in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Wosulin 7030/PK-PD/HV/FDA/10/3
Record Dates: First submitted 2011-05-20; First posted 2011-05-23 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wosulin 70/30 (Experimental): Wosulin 70N /30R is a recombinant Human Insulin with 30 % Regular Insulin Human Neutral and 70% Isophane Insulin, 600 nmol/ml, 100 IU/ml.
  Interventions: Biological: 30% Regular Insulin Human Neutral and 70%Isophane Insulin
- Novolin 70/30 (Active Comparator): Novolin 70/30 is a Recombinant Human Insulin with 70% NPH, Human Insulin Isophane Suspension and 30% Regular, Human Insulin Injection
  Interventions: Biological: Novolin 70/30

INTERVENTIONS:
Biological: 30% Regular Insulin Human Neutral and 70%Isophane Insulin — Total Dose per subject is 0.4 IU/Kg given subcutaneously.
  Arms: Wosulin 70/30
Biological: Novolin 70/30 — Total Dose per subject is 0.4IU/Kg given Subcutaneously.
  Arms: Novolin 70/30

SUMMARY:
The aim of this trial is to demonstrate bioequivalence of Wosulin 70/30 to Novolin® 70/30 with regard to its total and to its maximum serum insulin concentrations.

DETAILED DESCRIPTION:
The purpose of this study is is to test for bioequivalence based on AUC0-24h and Cmax between Wosulin 70N/30R and Novolin 70/30.The study also compares the pharmacokinetic and pharmacodynamic profiles as well as assessing safety and local tolerability of the two insulin preparations in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subject.
2. Age ≥ 18 and ≤ 45 years.
3. Considered generally healthy upon completion of medical history, physical examination and biochemical investigations as judged by the Investigator.
4. Body Mass Index (BMI) between 18.0 and 27.0 kg/m2, inclusive.
5. Non-smoker, defined as no nicotine consumption for at least one year.
6. Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.).

Exclusion Criteria:

1. Previous participation in this trial or other clinical trials within the last 30 days.
2. Pregnant, breast-feeding or intention of becoming pregnant or not using adequate contraceptive measures (defined as intrauterine device (IUD) that has been in place for at least 3 months, double barrier contraception, sterilization or abstinence, or oral contraceptive pill, which should have been taken without difficulty for at least 3 months, or an approved hormonal implant).
3. Clinically significant abnormal haematology or biochemistry screening tests, as judged by the Investigator. In particular, subjects with elevated liver enzymes (AST or ALT > 2 times the upper limit of normal) or impaired renal function (elevated serum creatinine values above the upper limit of normal) or fasting glucose at screening outside the range of 70-99 mg/dl will not be allowed to enter the trial.
4. Any serious systemic infectious disease during the four weeks prior to the first dose of test drug, as judged by the Investigator.
5. History of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose risk in administering the trial drug to the subject. In particular, subjects with significant cardiovascular disease, anemia (haemoglobin below the lower limit of normal) or hemoglobinopathy will not be allowed to enter the trial.
6. History of alcohol or drug abuse in the past five years.
7. Any positive test for drugs of abuse and /or alcohol at screening.
8. Hepatitis B or C or HIV positive.
9. Use of prescription drugs within 3 weeks preceding the first dosing of insulin, except for oral contraceptives/hormonal implants.
10. Treatment with any insulin product in the past.
11. Use of non-prescription drugs, except routine vitamins, within 2 weeks prior to the first dose of the test drug. Occasional use of acetaminophen is permitted.
12. Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation.
13. Blood donation of more than 500 ml within the last 12 weeks.
14. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
15. Known or suspected allergy to trial product or related products

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Mean AUC0-24h and Cmax | Visit 2 and 3

SECONDARY OUTCOMES:
PK endpts: AUC0-4h, AUC0-6h, AUC0-12h, AUC6-12h, AUC6-24h,tmax,and elimination rate constant. PD endpoints: AUCGIR0-4h, AUCGIR0-6h, AUCGIR0-12h,AUCGIR0-24h, AUCGIR6-12h, AUCGIR6-24h, GIRmax and tGIRmax Safety : AEs,haematology,biochem,phy exam | Visit 2,3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Marcus Hompesch, Study Director — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States